CLINICAL TRIAL: NCT02601469
Title: An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Maximal Use Treatment With DSXS (Taro Pharmaceuticals U.S.A., Inc.) in Patients With Plaque Psoriasis.
Brief Title: Study to Assess the Potential for Adrenal Suppression Following Treatment With DSXS in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSXS 1503
Record Dates: First submitted 2015-11-01; First posted 2015-11-10 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DSXS1503 (Experimental): administered twice daily for 28 days in patients with moderate to severe plaque psoriasis.
  Interventions: Drug: DSXS

INTERVENTIONS:
Drug: DSXS — twice daily for 28 days
  Other Names: Active

SUMMARY:
An open label, safety study to assess the potential for adrenal suppression following maximal use treatment with DSXS administered twice daily for 28 days in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
1. The objective of this study is to evaluate the potential of DSXS to suppress HPA axis function in patients with moderate to severe plaque psoriasis
2. To evaluate the efficacy parameters, pharmacokinetics and adverse event (AE) profile of DSXS

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of plaque psoriasis, patients 2-17 years of age with ≥ 10% BSA affected and patients age 18 years of age or older with ≥ 20% BSA affected
2. Investigator Global Assessment (IGA) score of 3 (moderate) or 4 (severe) at baseline for the overall disease severity.
3. Results from a cortisol response test that are considered normal and show no evidence of any abnormal HPA function or adrenal response

Exclusion Criteria:

1. Patients under 2 years of age.
2. Investigator Global Assessment (IGA) of less than 3 (moderate) or greater than 4 (severe) at baseline.
3. Current diagnosis of types of psoriasis other than stable plaque psoriasis (i.e., erythrodermic, exfoliative or pustular psoriasis).
4. Results from a cortisol response test that show evidence of any abnormal HPA function or adrenal response

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DSXS1503 Cohort 1: Administered twice daily for 28 days in patients with moderate to severe plaque psoriasis, age 19 years and older.
  DSXS: twice daily for 28 days
- DSXS1503 Cohort 2: Administered twice daily for 28 days in patients with moderate to severe plaque psoriasis, age 16-18 years of age.
  DSXS: twice daily for 28 days
Period: Overall Study
Arm/Group | DSXS1503 Cohort 1 | DSXS1503 Cohort 2
Started | 25 | 1
Completed | 24 | 1
Not Completed | 1 | 0
Not completed — Enrolled in Error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSXS1503 Cohort 1 | DSXS1503 Cohort 2 | Total
Number analyzed (Participants) | 25 | 1 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.72 (12.90) | 17.00 | 55.19 (14.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 1 | 11
  Male | 15 | 0 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 1 | 26
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 24 | 1 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Total BSA [Mean (Standard Deviation); unit: meters squared] | 2.11 (0.30) | 1.83 | 2.10 (0.30)
Baseline IGA [Count of Participants; unit: Participants]
  Clear | 0 | 0 | 0
  Minimal | 0 | 0 | 0
  Mild | 0 | 0 | 0
  Moderate | 20 | 1 | 21
  Severe | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HPA Axis Suppression
Description: Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the absence or presence of adrenal suppression at the end of treatment. HPA Axis suppression is defined as a 30 minute post CortrosynTM injection level cortisol level of ≤ 18 mcg/100ml.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS1503 Cohort 1 | DSXS1503 Cohort 2
Number analyzed (Participants) | 24 | 1
Participants
  Yes | 3 | 0
  No | 21 | 1

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Arm/Group | DSXS1503 Cohort 1 | DSXS1503 Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/1
Other Adverse Events (participants affected / at risk) | 7/25 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSXS1503 Cohort 1 (N=25) | DSXS1503 Cohort 2 (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
ACTH stimulation test abnormal (Investigations) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes